CLINICAL TRIAL: NCT05619562
Title: Clinical Significance of Circulating Tumour Cells in Resectable Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Responsible Party: Principal Investigator, Marian Hajduch, M.D., Ph.D., IMTM director, The Institute of Molecular and Translational Medicine, Czech Republic
Other Study IDs: NS10285
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Non Small Cell Lung Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA from plasma blood samples. DNA and RNA from nucleated blood cells. DNA and RNA from tumour tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Device for CTC/DTC detection — The CTCs/DTCs will be detected and counted in peripheral blood, tumour draining blood and bone marrow samples.

SUMMARY:
To determine whether the presence of circulating/disseminated tumour cells (CTCs/DTCs) in the blood and bone marrow of the resectable lung cancer (NSCLC) patients is a negative prognostic factor, and to find correlations with other clinical/pathological disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

Non-small cell lung cancer, non-metastatic

Exclusion Criteria:

Prior neoadjuvant chemoradiotherapy Prior lung cancer Cancer duplicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed non-metastatic NSCLC undergoing radical surgery with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
CEA, EGFR, LunX, c-met and EpCAM mRNA positive circulating tumour cells in lung cancer patients | 30 days
  The absolute gene expression of CEA, EGFR, LunX, c-met and EpCAM mRNA positive circulating tumour cells(CTCs) isolated from peripheral blood, tumour draining blood and bone marrow samples of lung cancer patients will be measured using real-time RT-PCR method. The gene expression will be normalized per microgram of total mRNA.

SECONDARY OUTCOMES:
Cancer specific survival in CTC positive NSCLC patients | 5 years
  The cancer specific survival, overall survival and disease free survival will be measured from the time of diagnosis to the time of event. Two groups of patients will be compared:
  A: Patients with the presence of CTCs in peripheral blood, tumour draining blood and bone marrow before NSCLC surgery as described in primary outcome measure.
  B: Patients with the absence e of CTCs in peripheral blood, tumour draining blood and bone marrow before NSCLC surgery as described in primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD, PhD, Study Director — Institute of Molecular and Translational Medicine, Faculty of Medicine and Dentistry, Palacky University
Locations (1):
- University Hospital Olomouc, Olomouc, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: No
The anonymized metadata will be publicly available after publishing the results.